CLINICAL TRIAL: NCT04936633
Title: Efficacy of Remote Intervention by Medical Staff Based on a Cloud System of Continuous Glucose Monitoring Data in Patients With Insulin-dependent Diabetes Using a Flash Sensor-based Glucose Monitoring (FSGM)
Brief Title: Efficacy of FSGM Cloud-based Remote Intervention for Insulin-dEpendent Diabetic Patients (FRIEND)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Young Shin Song (Other)
Responsible Party: Sponsor-Investigator, Young Shin Song, A ssistant Professor, CHA University
Organization: CHA University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-03-032-001
Record Dates: First submitted 2021-05-24; First posted 2021-06-23 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Remote intervention; Flash sensor-based glucose monitoring; Type 1 diabetes mellitus; Insulin-dependent diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention by medical staff (No Intervention): The patients who start FSGM and receive general education on FSGM only.
- Intervention by medical staff based on a cloud system (Experimental): The patients who start FSGM and receive general education on FSGM and remote intervention based on a cloud system.
  Interventions: Other: Intervention by medical staff based on a cloud system

INTERVENTIONS:
Other: Intervention by medical staff based on a cloud system — Remote intervention by medical staff (between Visit 1 and Visit 2; Week 2, 4, 6, 8, 10) : analyzing continuous glucose monitoring data for last two weeks in the cloud system
  - Intervention contents
  1. Diet, exercise pattern
  2. Causes of hypoglycemia
  3. Causes of hyperglycemia
  4. Causes of glycemic variability
  5. Counseling for improvement plans for the cause
  6. Counseling to strengthen lifestyle modification
  7. Counseling for insulin administration
  8. Counseling for Insulin dose adjustment (adjusted dose)
  9. Counseling for how to use a FSGM
  Arms: Intervention by medical staff based on a cloud system

SUMMARY:
To investigate the efficacy of remote intervention by medical staff based on a cloud system of continuous glucose monitoring data in patients with insulin-dependent diabetes using flash sensor-based glucose monitoring (FSGM).

DETAILED DESCRIPTION:
* Previous studies have been reported on the efficacy of CGM or FSGM and education on glucose control in insulin-dependent diabetes patients.
* This study aims to investigate whether it is more effective to receive remote intervention by medical staff based on a cloud system, than only to use FSGM and receive general education on FSGM.
* Trial design : parallel group, allocation ratio 1:1, a superiority study design

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 19 to 75 years old
* Patients with type 1 diabetes
* Patients on multiple daily insulin-injection or continuous subcutaneous insulin infusion therapy for more than 1 year
* Patients with HbA1c ≥ 7.0% at screening
* Patients willing to use a FSGM system
* Patients with informed consent

Exclusion Criteria:

* Gestational diabetes patients
* Patients within 1 year of diabetic diagnosis
* Patients taking drugs for severe cognitive impairment or psychiatric problems
* Patients who received oral or parenteral corticosteroid therapy for more than 7 consecutive days within 1 month before screening test
* Patients with severe infection, before and after surgery, and severe trauma
* Patients on dialysis at the end of renal failure
* Patients who have a history of substance abuse or alcoholism within 12 weeks through patient history taking, diagnosis records, and past treatment records
* Pregnant or lactating women
* Participating in other clinical trials under R&D other than this clinical trial, or if other clinical trial drugs are administered within 4 weeks before the trial
* Patients who are using a CGMS/FSGM or who have been using it within 12 weeks

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in glycemic control measured by HbA1c | 3 months
  Difference between baseline HbA1c and follow-up HbA1c

SECONDARY OUTCOMES:
Changes in the time in range | 3 months
  Difference in the duration of glucose values between 70 mg/dL and 180 mg/dL between baseline and the 3-month follow-up
Changes in the duration of hyperglycemic episodes | 3 months
  Difference in the duration of hyperglycemic glucose values (>180, 250 mg/dL) (baseline vs. follow-up)
Changes in the duration of hypoglycemic episodes | 3 months
  Difference in the duration of hypoglycemic glucose values (<70, 54 mg/dL) (baseline vs. follow-up)
Changes in hypoglycemic episodes | 3 months
  Difference between the frequency of hypoglycemic glucose values (<70, 54 mg/dL) (baseline vs. follow-up)
Changes in the mean glucose values | 3 months
  Difference in the mean glucose values (baseline vs. follow-up)
Changes in the frequency of use of trend arrows | 3 months
  Difference in the frequency of use of trend arrows (baseline vs. follow-up)
Changes in the mean number of scans | 3 months
  Difference in the mean number of scans per day (baseline vs. follow-up)
Changes in the insulin dose | 3 months
  Difference in the insulin dose (baseline vs. follow-up)
Changes in the lipid parameter | 3 months
  Difference in the levels of total cholesterol, triglycerides, HDL cholesterol, LDL cholesterol (baseline vs. follow-up)
Changes in blood pressure | 3 months
  Difference in systolic blood pressure and diastolic blood pressure (baseline vs. follow-up)
Changes in body weight | 3 months
  Difference in body weight (baseline vs. follow-up)
Lifestyle changes in diet | 3 months
  Difference in the average number of meals and snacks per day (baseline vs. follow-up)
Lifestyle changes in the number of exercises | 3 months
  Difference in the average number of exercises per week (baseline vs. follow-up)
Lifestyle changes in the duration of exercises | 3 months
  Difference in the average duration of exercises per week (baseline vs. follow-up)
Changes in the patient absolute satisfaction with treatment assessed by questionnaires | 3 months
  Difference in Diabetes Treatment Satisfaction Questionnaire Status (DTSQs) scores (baseline vs. follow-up)
Changes in the patient relative satisfaction with treatment assessed by questionnaires | 3 months
  Difference in Diabetes Treatment Satisfaction Questionnaire Change (DTSQc) scores (baseline vs. follow-up)
Changes in depression assessed by questionnaires | 3 months
  Difference in Patient Health Questionnaire-9 (PHQ-9) scores (baseline vs. follow-up)
Changes in anxiety assessed by questionnaires | 3 months
  Difference in General Anxiety Disorder-7 (GAD-7) scores (baseline vs. follow-up)

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Laffel LM, Kanapka LG, Beck RW, Bergamo K, Clements MA, Criego A, DeSalvo DJ, Goland R, Hood K, Liljenquist D, Messer LH, Monzavi R, Mouse TJ, Prahalad P, Sherr J, Simmons JH, Wadwa RP, Weinstock RS, Willi SM, Miller KM; CGM Intervention in Teens and Young Adults with T1D (CITY) Study Group; CDE10. Effect of Continuous Glucose Monitoring on Glycemic Control in Adolescents and Young Adults With Type 1 Diabetes: A Randomized Clinical Trial. JAMA. 2020 Jun 16;323(23):2388-2396. doi: 10.1001/jama.2020.6940. PMID 32543683
- [Background] Pratley RE, Kanapka LG, Rickels MR, Ahmann A, Aleppo G, Beck R, Bhargava A, Bode BW, Carlson A, Chaytor NS, Fox DS, Goland R, Hirsch IB, Kruger D, Kudva YC, Levy C, McGill JB, Peters A, Philipson L, Philis-Tsimikas A, Pop-Busui R, Shah VN, Thompson M, Vendrame F, Verdejo A, Weinstock RS, Young L, Miller KM; Wireless Innovation for Seniors With Diabetes Mellitus (WISDM) Study Group. Effect of Continuous Glucose Monitoring on Hypoglycemia in Older Adults With Type 1 Diabetes: A Randomized Clinical Trial. JAMA. 2020 Jun 16;323(23):2397-2406. doi: 10.1001/jama.2020.6928. PMID 32543682
- [Background] Hermanns N, Ehrmann D, Schipfer M, Kroger J, Haak T, Kulzer B. The impact of a structured education and treatment programme (FLASH) for people with diabetes using a flash sensor-based glucose monitoring system: Results of a randomized controlled trial. Diabetes Res Clin Pract. 2019 Apr;150:111-121. doi: 10.1016/j.diabres.2019.03.003. Epub 2019 Mar 4. PMID 30844467
- [Derived] Lee J, Lee MH, Park J, Kim KS, Kim SK, Cho YW, Han HW, Song YS. FGM-based remote intervention for adults with type 1 diabetes: The FRIEND randomized clinical trial. Front Endocrinol (Lausanne). 2022 Nov 25;13:1054697. doi: 10.3389/fendo.2022.1054697. eCollection 2022. PMID 36506077